CLINICAL TRIAL: NCT07325188
Title: Clinical Evaluation of a Novel Intraoperative Guidance System for Accurate Toric IOL Positioning in Cataract Surgery
Brief Title: HUD Surgical Guidance for Toric Alignment
Acronym: CG-Toric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gainesville Eye Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0104
Record Dates: First submitted 2025-12-04; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cataract and IOL Surgery
Keywords: Guidance; Toric IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Surgical guidance for Toric IOL alignment intraoperatively (Other): Interventional
  Interventions: Device: Cassini Guidance

INTERVENTIONS:
Device: Cassini Guidance — Cassini Guidance with HUD

SUMMARY:
This study aims to assess the accuracy of toric intraocular lens (IOL) alignment axes as calculated and displayed by a novel digital guidance system. In addition, it evaluates the time required to initiate surgical guidance and postoperative refractive astigmatism following toric IOL implantation.

This single-surgeon, single-site, prospective, non-invasive observational study evaluated the accuracy of toric IOL alignment axes calculated and displayed by the digital guidance system (Cassini Technologies, B.V.) in 100 eyes. The intraoperatively calculated alignment axes were compared to preoperative measurements to assess their accuracy (in degrees). Postoperative outcomes, including residual refractive astigmatism (diopters) and visual acuity (Snellen), were recorded at 1 month postoperatively.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing uncomplicated cataract surgery with toric IOL implantation,
* Eyes implanted with a toric IOL.

Exclusion criteria:

* Ocular comorbidity likely to impair postoperative visual acuities, or
* History of ocular trauma or zonular instability, or
* Previous refractive surgery, or
* Irregular corneal astigmatism or keratoconus, or
* Patients with physical or intellectual disabilities that may prevent reliable fixation or comprehension (e.g. Down's Syndrome, Parkinson's Disease), or
* Patients with unreliable biometry measurements, or
* Severe dry eye disease or ocular surface disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy (measured in degrees of arc) using the Cassini Guidance system for calculated alignment axis for toric IOL implantation. | Total completion up to 12 months
  Primary Endpoint:
  1. Accuracy of the calculated alignment axis (degrees of arc = angular degrees)
  * Definition: The angular difference between the alignment axis for toric IOLs as determined with the CGS and the intended alignment axis as determined with the Cassini Ambient.
  * Thresholds of interest: ≤3°, ≤5°, ≤10°, >10°.
  * Justification: Misalignment greater than 10° results in a clinically significant loss of toric correction (approximately 33%) (Quesada et al., 2022; Hu, 2023), making this a meaningful accuracy benchmark.

SECONDARY OUTCOMES:
Time efficiency (measured in seconds) of the Cassini Guidance System in eyes undergoing cataract surgery with toric IOL implantation. | Total completion up to 12 months
  Secondary Endpoint:
  1. The time (measured in seconds) required to initiate (0 seconds) and finish (x seconds) surgical guidance using the Cassini Guidance System in 100 eyes undergoing toric IOL implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- North Georgia Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao L, Jia S, Yang X, Li M, Yu X, Zhao P, Bai H. Image-Guided Marking versus Manual Marking in Phacoemulsification with Toric Intraocular Lens (IOL) Implantation: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Semin Ophthalmol. 2024 Jan;39(1):60-65. doi: 10.1080/08820538.2023.2231575. Epub 2023 Jul 3. PMID 37400160